CLINICAL TRIAL: NCT02112084
Title: Enhancing End-of-Life and Bereavement Outcomes Among Cancer Caregivers: Individualized Dual Process Intervention for Bereaved Partners After Cancer Death
Brief Title: An Individualized Grief Intervention for Spouses of Cancer Patients After the Patient's Death
Acronym: DPM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kathleen Mooney, Principal Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 33122-DPM; 1P01CA138317 (NIH)
Record Dates: First submitted 2014-04-02; First posted 2014-04-11 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-02

CONDITIONS: Bereavement; Death; Cancer
MeSH Terms: conditions — Death; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (No Intervention): Usual care participants do not receive an intervention.
- Individualized DPM (Experimental): Individualized DPM
  Interventions: Behavioral: Individualized DPM

INTERVENTIONS:
Behavioral: Individualized DPM — The intervention includes 7 LO phone sessions and 7 RO home visits provided by trained interventionists. The primary focus of the LO phone conversations will be on grief work issues, daily functioning, and emotional support. The calls will provide an opportunity to discuss how grief could be interfering with their daily functioning, dealing with grief-related feelings- emotions they are experiencing, the frustrations associated with taking on new responsibilities while still trying to meet their own needs, critical time periods like anniversaries and holidays, unfinished business, coping strategies, including using humor, and having realistic expectations about the bereavement process. The RO home visits will be based specifically on the bereaved partners' skill and knowledge needs.
  Arms: Individualized DPM

SUMMARY:
Individuals providing end-of-life caregiving to partners with terminal cancer often begin the bereavement process before the patient dies and with additional sources of stress. We know that grief for these partners can be long-term and impact virtually every aspect of their lives. This project will test the effectiveness of a new promising intervention that uses a dual process model (DPM) which focuses both on loss orientation (emotional loss and grief (referred to as LO)) and restoration orientation (learning new tasks of living that may have been the primary responsibility of the spouse who has died (referred to as RO tasks)).

DETAILED DESCRIPTION:
The past emphasis on only the psycho-emotional features of loss has resulted in a lack of attention to the restoration-focused adaptation. Middle-aged and older bereaved persons, including those who previously provided care for a terminally ill spouse or partner, are confronted with unfamiliar daily demands. Even though death due to a terminal illness like cancer may be anticipated, the surviving spouse/partner may be so involved in caring for the dying person and consumed by the emotional distress that accompanies it, there is little time or energy to plan for the changes, some of which are unforeseen prior to the loss. This gap in abilities suggests a need for intervention strategies that improve skills such as mastering tasks of daily living, engaging in self-care behaviors, and functioning socially as a single or uncoupled person in society. One of the major findings in our previous research was the strong association between competencies in tasks of daily living and more favorable adjustments to psycho-emotional aspects of grief.

Some tasks of daily living may have been the primary responsibility of the deceased person. If these skills are not acquired during bereavement, the health, functioning, autonomy and overall quality of life of the bereaved could be adversely affected. Furthermore, the inability to accomplish these tasks interferes with the emotion-focused energy the bereaved need to direct toward the loss itself. Effectively coping with the secondary stress associated with these new challenges reduces the emotional disruption of bereavement. As new skills are gained, the bereaved feel more confident to meet future challenges in their daily lives and some may experience personal growth as they venture into "previously uncharted territory" during a time of transformation independent of their deceased spouses/partners.

While some of the RO challenges are practical, others have health implications (some have both). Self-care behaviors are often partnered activities among couples and the partner's death frequently disrupts these behavioral patterns or interferes with the ability to engage in new ones. The importance for bereaved persons to care for themselves while still addressing the need to grieve represents another set of secondary stressors requiring RO coping strategies. Also, those who more effectively engage in self-care could conceivably be in a better position to address the negative emotional effects of the loss. An important feature of RO is the adaptation to new roles and identities and establishing new relationships and maintaining social connectedness. Older and middle aged bereaved spouses/partners prefer to maintain the meaningful relationships and activities they have had throughout their lives but they also want to learn ways to access services and programs more effectively and how to maximize opportunities to meet and socialize with others. Activities can include inexpensive entertainment and leisure options, safe places to go to socialize with others, and volunteering opportunities to help others so they can remain socially connected and function more effectively and comfortably as a single person. These activities provide potential linkages to the service network and opportunities for time away from grief itself.

The overall intent of the I-DPM intervention is to more effectively stimulate both LO and RO coping processes as well as the oscillation between them than what would otherwise occur without an exposure to such a treatment. At best the usual care hospice caregivers receive after the death of the patient is primarily LO focused as well as infrequent. We hypothesize that those who receive the I-DPM intervention will show greater improvements over time in bereavement outcomes largely because the intervention content will stimulate both LO and RO processes - the telephone support will focus primarily on LO coping while the home visits are intended to address RO issues causing the most concern for the bereaved. In our earlier work we documented that LO coping was directly related to grief, depression, bereavement coping self-efficacy, and loneliness, while RO coping was strongly associated with competencies and personal growth. RO coping, however, also was related to the aforementioned loss-oriented outcomes most likely because of the positive relationship between competencies and the psycho-emotional aspects of bereavement mentioned above and the confidence one can master new challenges along with the perception of growth that accompanies it.

To summarize, bereavement interventions that have traditionally focused on grief work and psycho-emotional outcomes have only been moderately effective, largely due to having a limited focus on emotional coping. Alternatively, an intervention that addresses RO in addition to LO as we are testing in the DPM intervention could provide a more promising solution by helping the bereaved develop skills specific to practical daily challenges as well as the emotional disruption and upset that permeate bereavement.

ELIGIBILITY:
Inclusion Criteria:

* Spouse/Partner of patient with a cancer diagnosis who received hospice care in their home by one of the participating hospice programs
* Lived in the home with the patient
* English speaking and writing
* cognitively and physically able to use the phone unassisted, complete questionnaires, and participate in the DPM intervention
* Access to a telephone
* Intends to reside in an area where the intervention will be offered for the time it takes to deliver the intervention (14 weeks from the start of the intervention).

No Exclusion Criteria:

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2010-05; Primary Completion 2016-03 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
DPM Coping Processes: Loss- and Restoration- Orientation and Oscillation | up to 14 months post patient death
  Features of the DPM will be measured using the Inventory of Daily Widowed Life (IDWL) which consists of 22 Likert-format items that inquire into how much time during the past week the respondents spend on loss-orientation (e.g., "Thinking about how much I miss my spouse;" "Feeling a bond with my spouse") and restoration-oriented activities (e. g., "Finding ways to keep busy or occupied;" "Took some time away from grieving for my spouse"). At the end of the 22 IDWL items are several additional questions we developed to measure important dimensions of the oscillation between LO and RO. These features assess oscillation awareness, frequency, and control (each measured on a 5-point Likert scale) and oscillation intent is measured by an open-ended item that asks, "When I go back and forth between dealing with these two issues (grief-related emotions vs. new responsibilities, activities and time away from grieving), I usually do it because __.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen H Mooney, PhD, Principal Investigator — University of Utah; Michael Caserta, PhD, Study Chair — University of Utah; Dale Lund, PhD, Study Chair — California State University, San Bernardino
Locations (1):
- University of Utah College of Nursing, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No